CLINICAL TRIAL: NCT05803408
Title: A Randomized Controlled Trial to Evaluate Effect of Late vs Early Introduction of Gluten-free Oats on Symptomatic, Serologic and Disease Activity in Patients With Newly Diagnosed Celiac Disease.
Brief Title: RCT: Effect of Late vs Early Introduction of Gluten-free Oats on Patients With Newly Diagnosed Celiac Disease.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Maria Ines Pinto Sanchez, Associate Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 15964
Record Dates: First submitted 2023-01-24; First posted 2023-04-07 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Celiac Disease; Gluten Sensitivity; Gluten Allergy; Gluten Enteropathy
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early introduction of gluten free oats (Experimental): Early introduction of oats (starting GF oats immediately after the diagnosis, within 3 months)
  Interventions: Other: gluten-free oats
- Late introduction of gluten free oats (Active Comparator): Late introduction of oats (starting GF oats 6 months after diagnosis of celiac disease)
  Interventions: Other: gluten-free oats

INTERVENTIONS:
Other: gluten-free oats — Early vs late introduction of gluten free oats

SUMMARY:
The investigators are conducting a pilot study to investigate the impact of late compared to early introduction of gluten-free oats on gut symptoms, nutrition status, celiac activity and quality of life in patients with a recent diagnosis of celiac disease. Pilot study means that it will recruit a low number of participants to see if it is possible to perform the study, and to estimate how many participants will be needed for the large study. The study will collect information through questionnaires that assess gut symptoms, quality of life, mood changes and dietary patterns. Moreover, the study will collect data on tests done during clinic visits to check the status of patients' celiac markers and nutritional status (such as vitamins and minerals). Physical exam will also take place, and include measurement of weight, BMI and body composition in a 3D scanner. The dietitian will analyze patients' diet at each visit during the study period. Given the lack of evidence on timing of introduction of gluten-free oats for patients with a recent celiac diagnosis, and the potential risks of limiting oats in a gluten-free diet, the results will hopefully lead to better understanding of whether one strategy has a benefit over the other.

DETAILED DESCRIPTION:
Celiac disease (CeD) is a chronic inflammatory condition triggered by gluten in genetically predisposed individuals, manifesting with both intestinal and extra-intestinal symptoms. There is a relatively high prevalence of CeD in Western populations of around 1%. People with CeD have adverse immune-mediated reactions to gluten, which is the most abundant protein in many cereal grains, including wheat, rye, and barley. Currently, the only available treatment for CeD is a gluten-free diet (GFD). Gluten-free products are defined as containing less than 20 ppm of gluten, an international standard set by Codex Alimentarius Commission based on scientific data.

Oats are safe for most people with CeD, provided they are pure and uncontaminated with gluten. A small proportion of patients will react to avenin, the protein contained in oats, but this does not lead to intestinal inflammation. However, oats, including some brands labelled as gluten-free, are often contaminated with gluten, most notably from cross-contamination with wheat and barley due to agricultural practices. Furthermore, many patients remain symptomatic despite adhering to a GFD for different reasons, and concerns have been raised over whether continue eating oats to a GFD may contribute to persisting symptoms. For this reason, some experts in CeD recommend to delay the introduction of oats until 6 months after the diagnosis as part of a stabilization phase, after which the CeD is under better control and TTG autoantibody levels have decreased. However, there is no evidence this approach has any benefit over permitting the intake of GF oats from the time of diagnosis.

A GFD is restrictive and has been associated with nutritional deficiencies. Oats are highly nutritious and possess additional health benefits. They are an excellent source of macro- and micro-nutrients, including B complex vitamins, minerals, and heart-healthy soluble dietary fiber. These nutrients are essential in prevention of many chronic diseases such as diabetes and reducing cardiovascular risk factors. In addition, preliminary research suggests a benefit of oats on the gut microbiome.

Considering how rarely CeD patients react to oats and the numerous benefits of oats for nutrition and overall health, the delayed introduction of oats into the GFD, provided they are certified GF, has come under scrutiny. Given the lack of evidence that a delayed introduction of oats is beneficial for CeD patients and the potential risks of limiting oats in a GFD, there is an unmet need to understand the benefits of one approach over the other to provide recommendations for clinical practice.

This study proposes a pilot randomized controlled trial (RCT) to investigate the impact of late compared to early introduction of oats on gastrointestinal symptoms, nutritional status, disease activity and quality of life in patients with a recent diagnosis of CeD. The results of this study will provide the basis to plan an adequately powered RCT, and the results of the study will be highly relevant to guide recommendations in clinical practice on when oats should be introduced to patients with a CeD diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Recent diagnosis of CeD (within 3 months of starting a GFD) based on specific CeD serology (elevated anti-tissue transglutaminase IgA, deaminated gliadin peptides IgG or anti-endomysial antibodies IgA) and confirmed by duodenal biopsies showing villous atrophy (Marsh 3a or greater). The allowance of 3 months is related to 1) the time lag between tTG and confirmatory EGD testing in clinical practice and 2) the time lag between diagnosis and dietitian assessment, which will increase likelihood of achieving a strict GFD.

Exclusion Criteria:

1. Have already removed oats from the diet;
2. History of allergic reaction to oats
3. Prior assessment and education by RD on GFD
4. Unwillingness or inability to commit to study procedures *Patients receiving antibiotics or probiotics within a month will be allowed to participate, however, this will be documented for future microbiota analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Better symptom control | 3-6 months
  To assess the impact of late (after 6 months) vs early (immediate) introduction of gluten-free oats as part of a gluten-free diet on achieving better symptom control (change in Celiac Disease Gastrointestinal Symptom Rating Scale scores; range 15-115; lower the score, the better the outcome) at 3- and 6-month follow-up
tTG antibody levels | 6 months
  To assess the impact of late (after 6 months) vs early (immediate) introduction of gluten-free oats as part of a gluten-free diet on achieving:
  Change in tTG antibody levels at 6-month follow-up
improvement of nutritional status | 6 months
  To assess the impact of late (after 6 months) vs early (immediate) introduction of gluten-free oats as part of a gluten-free diet on achieving:
  improvement of nutritional status (reduce % body fat mass)
improvement in quality of life (change in Celiac Disease Quality of Life scores) | 3-6 months
  To assess the impact of late (after 6 months) vs early (immediate) introduction of gluten-free oats as part of a gluten-free diet on achieving:
  improvement in quality of life (change in Celiac Disease Quality of Life scores, 20-100, lower the score better the outcome) at 3- and 6-month follow-up
Food insecurity | 6 months
  Food insecurity will be assessed through Household Food Security Survey Module (HFSSM)

CONTACTS AND LOCATIONS:
Overall Officials: Jedid-Jah Blom, RD, Study Director — Hamilton Health Sciences Corporation
Locations (1):
- McMaster University Medical Center, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No